CLINICAL TRIAL: NCT00692991
Title: Microvascular Obstruction by Contrast-enhanced MRI Following Percutaneous Coronary Interventions
Brief Title: Using Magnetic Resonance Imaging to Evaluate Heart Vessel Function After Angioplasty or Stent Placement Procedures
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Katherine C. Wu, Associate Professor of Medicine, Johns Hopkins University
Other Study IDs: 566; K23HL004444-01 (NIH)
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2013-02

CONDITIONS: Myocardial Infarction; Angina, Unstable; Cardiomyopathy, Hypertrophic
Keywords: Microvascular Obstruction; Cardiac MRI; Alcohol Ablation; Diagnostic PCI
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: People undergoing percutaneous coronary interventions.

SUMMARY:
Coronary artery disease (CAD) is caused by a narrowing of the blood vessels that supply blood and oxygen to the heart. Balloon angioplasty and stent placement are two treatment options for people with reduced heart function caused by CAD. This study will use magnetic resonance imaging (MRI) procedures to evaluate heart function over time in people with CAD who have undergone a balloon angioplasty or stent placement procedure.

DETAILED DESCRIPTION:
CAD is the most common type of heart disease in the United States. It occurs when the arteries that supply blood to the heart become hardened and narrowed because of a build-up of cholesterol and plaque on the inner walls of the arteries. Over time, less blood is able to flow through the arteries, depriving the heart of the blood and oxygen it needs. If left untreated, CAD can lead to heart failure, heart attack, and arrhythmias. Someone with plaque build-up may undergo a percutaneous coronary intervention (PCI) to unblock the narrowed arteries and increase blood flow. PCI encompasses a variety of procedures, including balloon angioplasty and stent placement. In balloon angioplasty, a small balloon is inserted into the heart artery and then inflated. This pushes the plaque against the artery walls and widens the artery. Stents are wire mesh tubes that are permanently implanted in the artery to keep it propped open. Although balloon angioplasty and stent placement procedures open up blockages in the large vessels of the heart, the tiny vessels of the heart may become blocked after these procedures, which may affect how the heart heals. This study will use MRI to examine heart function in people who have undergone PCI procedures. Study researchers will attempt to define how often blockages of the tiny vessels occur after PCI procedures, the factors that lead to the blockages, and how often blockages affect healing of the heart.

This study will enroll people who are undergoing a PCI procedure. Participants will undergo an MRI scan of the heart before and after the PCI procedure. During the 72 hours after the procedure, electrocardiogram (EKG) will be used to monitor heart electrical activity. At a study visit 10 days after the PCI procedure and at a follow-up visit 6 to 12 months later, participants will undergo an MRI, EKG, and blood collection. Study staff will call participants every 6 months for 5 years to collect medical information.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing diagnostic coronary angiography
* Undergoing percutaneous coronary intervention

Exclusion Criteria:

* Clinically unstable (i.e., demonstrates unstable cardiac rhythm or hemodynamics, supported on vasopressors or an intra-aortic balloon pump, and/or is actively ischemic) at the time of the MRI procedure
* Unable to undergo MRI procedure (e.g., has non-MRI compatible implanted metallic objects, including cardiac pacemakers or cerebral aneurysm clips that are not MRI compatible)
* Current glomerular filtration rate of less than 60mL/min/1.73m2
* Pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed on the cardiac catheterization schedule who are undergoing percutaneous coronary interventions.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 1999-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of microvascular obstruction by MRI in participants who may or may not have had an acute heart attack; coronary angiographic correlates of MRI microvascular obstruction | Measured during participant's initial and follow-up MRIs

SECONDARY OUTCOMES:
Relation of presence and extent of microvascular obstruction to clinical outcomes over 5 years | Measured every 6 months for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Wu, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Johns Hopkins Medical Institution, Baltimore, Maryland, United States

REFERENCES:
- [Background] Fernandes VR, Wu KC, Rosen BD, Schmidt A, Lardo AC, Osman N, Halperin HR, Tomaselli G, Berger R, Bluemke DA, Marban E, Lima JA. Enhanced infarct border zone function and altered mechanical activation predict inducibility of monomorphic ventricular tachycardia in patients with ischemic cardiomyopathy. Radiology. 2007 Dec;245(3):712-9. doi: 10.1148/radiol.2452061615. Epub 2007 Oct 2. PMID 17911537
- [Background] Rettmann DW, Saranathan M, Wu KC, Azevedo CF, Bluemke DA, Foo TK. High temporal resolution breathheld 3D FIESTA CINE imaging: validation of ventricular function in patients with chronic myocardial infarction. J Magn Reson Imaging. 2007 Jun;25(6):1141-6. doi: 10.1002/jmri.20923. PMID 17520725
- [Background] Murthy VL, Wu KC. Advances in cardiac MRI: The multi-ethnic study of atherosclerosis. Curr Cardiol Rep. 2007 Mar;9(1):43-4. No abstract available. PMID 17436456
- [Background] Murthy VL, Wu KC. Advances in cardiac MRI: The Dallas Heart Study. Curr Cardiol Rep. 2007 Mar;9(1):43. No abstract available. PMID 17436455
- [Background] Schmidt A, Azevedo CF, Cheng A, Gupta SN, Bluemke DA, Foo TK, Gerstenblith G, Weiss RG, Marban E, Tomaselli GF, Lima JA, Wu KC. Infarct tissue heterogeneity by magnetic resonance imaging identifies enhanced cardiac arrhythmia susceptibility in patients with left ventricular dysfunction. Circulation. 2007 Apr 17;115(15):2006-14. doi: 10.1161/CIRCULATIONAHA.106.653568. Epub 2007 Mar 26. PMID 17389270
- [Background] Azevedo CF, Amado LC, Kraitchman DL, Gerber BL, Edvardsen T, Osman NF, Rochitte CE, Wu KC, Lima JA. The effect of intra-aortic balloon counterpulsation on left ventricular functional recovery early after acute myocardial infarction: a randomized experimental magnetic resonance imaging study. Eur Heart J. 2005 Jun;26(12):1235-41. doi: 10.1093/eurheartj/ehi137. Epub 2005 Feb 16. PMID 15716282
- [Background] Kumbasar B, Wu KC, Kamel IR, Lima JA, Bluemke DA. Left ventricular true aneurysm: diagnosis of myocardial viability shown on MR imaging. AJR Am J Roentgenol. 2002 Aug;179(2):472-4. doi: 10.2214/ajr.179.2.1790472. No abstract available. PMID 12130455
- [Result] Heldman AW, Wu KC, Abraham TP, Cameron DE. Myectomy or alcohol septal ablation surgery and percutaneous intervention go another round. J Am Coll Cardiol. 2007 Jan 23;49(3):358-60. doi: 10.1016/j.jacc.2006.10.029. Epub 2007 Jan 4. No abstract available. PMID 17239718
- [Result] Luo AK, Wu KC. Imaging microvascular obstruction and its clinical significance following acute myocardial infarction. Heart Fail Rev. 2006 Dec;11(4):305-12. doi: 10.1007/s10741-006-0231-0. PMID 17131076
- [Result] Vogel-Claussen J, Rochitte CE, Wu KC, Kamel IR, Foo TK, Lima JA, Bluemke DA. Delayed enhancement MR imaging: utility in myocardial assessment. Radiographics. 2006 May-Jun;26(3):795-810. doi: 10.1148/rg.263055047. PMID 16702455
- [Result] Schmidt A, Wu KC. MRI assessment of myocardial viability. Semin Ultrasound CT MR. 2006 Feb;27(1):11-9. doi: 10.1053/j.sult.2005.11.001. PMID 16562568
- [Result] Wu KC. Assessment of non-st-segment elevation acute coronary syndromes with cardiac MRI. Curr Cardiol Rep. 2006 Feb;8(1):42-3. No abstract available. PMID 16507235
- [Result] Wu KC. Utility of cardiac MRI in the diagnosis of hypertrophic cardiomyopathy. Curr Cardiol Rep. 2006 Feb;8(1):41. No abstract available. PMID 16507234
- [Result] Lardo AC, Cordeiro MA, Silva C, Amado LC, George RT, Saliaris AP, Schuleri KH, Fernandes VR, Zviman M, Nazarian S, Halperin HR, Wu KC, Hare JM, Lima JA. Contrast-enhanced multidetector computed tomography viability imaging after myocardial infarction: characterization of myocyte death, microvascular obstruction, and chronic scar. Circulation. 2006 Jan 24;113(3):394-404. doi: 10.1161/CIRCULATIONAHA.105.521450. PMID 16432071
- [Result] Foo TK, Ho VB, Saranathan M, Cheng LQ, Sakuma H, Kraitchman DL, Wu KC, Bluemke DA. Feasibility of integrating high-spatial-resolution 3D breath-hold coronary MR angiography with myocardial perfusion and viability examinations. Radiology. 2005 Jun;235(3):1025-30. doi: 10.1148/radiol.2353040090. PMID 15914483
- [Result] Foo TK, Stanley DW, Castillo E, Rochitte CE, Wang Y, Lima JA, Bluemke DA, Wu KC. Myocardial viability: breath-hold 3D MR imaging of delayed hyperenhancement with variable sampling in time. Radiology. 2004 Mar;230(3):845-51. doi: 10.1148/radiol.2303021411. PMID 14990846
- [Result] Wu KC, Lima JA. Noninvasive imaging of myocardial viability: current techniques and future developments. Circ Res. 2003 Dec 12;93(12):1146-58. doi: 10.1161/01.RES.0000103863.40055.E8. PMID 14670830
- [Result] Wu KC. Myocardial perfusion imaging by magnetic resonance imaging. Curr Cardiol Rep. 2003 Jan;5(1):63-8. doi: 10.1007/s11886-003-0039-7. PMID 12493162
- [Result] Gerber BL, Garot J, Bluemke DA, Wu KC, Lima JA. Accuracy of contrast-enhanced magnetic resonance imaging in predicting improvement of regional myocardial function in patients after acute myocardial infarction. Circulation. 2002 Aug 27;106(9):1083-9. doi: 10.1161/01.cir.0000027818.15792.1e. PMID 12196333